CLINICAL TRIAL: NCT00792766
Title: Long Term Follow Up for RAD001 Therapy of Angiomyolipomata in Patients With Tuberous Sclerosis Complex and Sporadic Lymphangioleiomyomatosis
Brief Title: Long Term Follow Up for RAD001 Therapy of Angiomyolipomata in Patients With Tuberous Sclerosis (TSC) and Sporadic Lymphangioleiomyomatosis (LAM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC IRB# 2008-0333
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Tuberous Sclerosis; Angiolipoma
Keywords: Tuberous Sclerosis Complex (TSC); Angiolipoma; mTOR; Everolimus
MeSH Terms: conditions — Tuberous Sclerosis; Angiolipoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: everolimus (RAD001)

INTERVENTIONS:
Drug: everolimus (RAD001) — Subjects will resume the dosing regimen that they were receiving at the completion of the initial RAD001 study.
  Other Names: RAD001

SUMMARY:
This is an open label long term follow up study, open to those subjects who were previously enrolled in"RAD001 Therapy of Angiomyolipomata in Patients with Tuberous Sclerosis Complex and Sporadic Lymphangioleiomyomatosis", CCHMC IRB #2008-0812 and who meet the criteria for this long-term follow-up study.

The hypothesis is that the drug will inhibit the growth of the angiomyolipomas and possibly even cause regression.

DETAILED DESCRIPTION:
Tuberous sclerosis complex is a genetic disorder with a birth incidence of approximately one in six thousand. Angiomyolipomas occur in eighty percent of persons with TS, and in up to 60% of persons with LAM. They are fatty tumors that often occur in kidney or liver as well as other parts of the body. They can grow and cause damage to surrounding kidney tissue and even renal failure. They may also leak blood causing potentially life-threatening hemorrhage.

Laboratory studies have shown that RAD001 suppresses the chemical that cause tumors to grow in tuberous sclerosis and sporadic LAM. The use of RAD001 to treat angiomyolipomas in tuberous sclerosis or sporadic LAM is considered experimental.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have met all eligibility criteria for the initial RAD001 protocol (CCHMC IRB 2008-0812)
* Subjects with documented angiomyolipoma volume decrease from baseline measures at the end of 12 months on study drug of thirty percent or more during the initial RAD001 protocol OR subjects with less than thirty percent decrease in angiomyolipomas at the end of 12 months on study drug but with documented improvement, or stabilization, of baseline clinical status per physical, pulmonary function and/or laboratory examination at the end of 12 months on study drug that was not maintained during a period of 12 or more months off study drug.
* If female and of child-bearing potential, documentation of negative pregnancy test prior to start of study drug
* Creatinine <3 mg/dl, within 30 days prior to start of drug

Exclusion Criteria:

* Inability to complete the initial RAD001 protocol (CCHMC IRB # 2008-0812) due to toxicities requiring discontinuation of treatment.
* Demonstrated an increase in the size of the angiomyolipoma from baseline at the end of 12 months on study drug on the initial RAD001 study.
* Significant hematologic or hepatic abnormality (i.e. ALT and AST >2.5x ULN), serum albumin <3 g/dl, HCT <30%, platelets <75,000/cumm, adjusted absolute neutrophil count <1,000/cumm, total WBC <3,000/cumm).
* Continuous requirement for supplemental oxygen.
* Intercurrent infection at initiation of RAD001.
* Embolization of angiomyolipoma within one month; any other recent surgery (within 2 months of initiation of RAD001).
* Pregnant or lactating women or women who plan on becoming pregnant during the course of this study due to unknown effects of RAD001 on the fetus.
* Inadequate contraception (participants who are fertile must maintain adequate contraception throughout the trial and for three months after stopping the drug). Acceptable contraceptive measures include non estrogen-containing birth control contraceptive regimen (progestin based contraceptives), prior hysterectomy, tubal ligation, complete abstinence, barrier methods which include a cervical diaphragm and spermicidal jelly, IUD, or vasectomy in partner.
* Use of an investigational drug, including rapamycin, within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
RAD001 tolerance | Every three months while on study drug

SECONDARY OUTCOMES:
Angiomyolipoma volume reduction | Every year while on study drug

CONTACTS AND LOCATIONS:
Overall Officials: John Bissler, MD, Principal Investigator — LeBonheur Children's Hospital
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States